CLINICAL TRIAL: NCT03853252
Title: iPS Cells of Patients for Models of Retinal Dystrophies
Acronym: RETIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9366
Record Dates: First submitted 2019-02-22; First posted 2019-02-25 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Retinal Dystrophies
MeSH Terms: conditions — Retinal Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Skin biopsy (Other)
  Interventions: Other: Skin biopsy

INTERVENTIONS:
Other: Skin biopsy — Skin biopsy on a location preliminarily anesthetized Disinfection protocol Combined required blood tests (HIV, Hepatitis B)

SUMMARY:
The investigators are focused on inherited retinal dystrophies with an aim to further understand disease pathophysiology and to elaborate novel treatments, as, to date, there is no effective treatment to prevent blindness.

The main goal of this study is to generate human cellular models of healthy and disease retinas and perform studies to evaluate the efficiency of gene therapy approaches for different diseases.

Skin biopsies of volunteers are cultured to isolate fibroblasts that are then reprogrammed into iPS cells. Healthy and disease-specific iPS cells are then differentiated into retinal models.

This study should help to elucidate disease pathways and to provide proof-of-concept for various therapeutic approaches.

ELIGIBILITY:
Inclusion criteria :

* Signed informed consent and
* Choroideremia :

  * Males
  * CHM mutation
  * With multimodal Imaging anomalies in line with CHM
* All other presumed inherited retinal dystrophies with bilateral and symmetrical involvement with identified mutations in one of the Retnet gene
* All presumed inherited optic neuropathy with bilateral and symmetrical involvement with identified mutations
* And in all cases or pattern

  * Age from 5 to 70
  * with appropriate health insurance

Exclusion criteria :

* Patient under tutorship or curatorship

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-11-03 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
number of human cell models obtained | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- CNMR Maolya, Genetic Sensory Diseases, Montpellier, Occitanie, France

IPD SHARING:
Plan to Share IPD: No